CLINICAL TRIAL: NCT06169826
Title: Histidine Oral Supplementation as a Therapeutic Modality for Alzheimer's Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: withdrawn by the PI
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00093174
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Histidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control
  Interventions: Other: Control
- Treatment-Histidine (Active Comparator): Treatment-Histidine
  Interventions: Drug: l-Histidine

INTERVENTIONS:
Drug: l-Histidine — In the outpatient setting, one chewable tablet multivitamin (Zn and folic acid containing) plus a titrated dosing of L-histidine powder or capsules starting at 2g consumed before noon escalating every 2 weeks up to 4, 6, then 8 g per day as tolerated for up to 3 months.
  Arms: Treatment-Histidine
Other: Control — Control
  Arms: Control

SUMMARY:
Oral supplementation of histidine in patients with cognitive dysfunction should increase brain anserine, carnosine and histamine levels which will result in improved cognition via numerous proven in vivo mechanisms including increasing blood flow, neurogenesis, angiogenesis, activation of histaminergic neural pathways and autophagy of beta-amyloid protein, which is pathognomonic for Alzheimer's disease.

Randomized into one of 2 arms to receive Histidine or placebo to take for up to 3 months. Baseline evaluation and followup evaluation at 3 months postop.

DETAILED DESCRIPTION:
The patients will be offered enrollment by sequential measures with odd numbers placed into the Control Group and even numbers in the Treatment Arm. One hundred patients will be enrolled in each arm. Study medications will be initiated in the outpatient setting following informed consent, enrollment and baseline lab evaluation. Scheduled clinic visits at 3 months and 1 year from date of enrollment will be used to re-assess performance via repeat cognitive testing. Lab evaluation of CBC, CMP, histidine and histamine levels will occur at baseline and the 3 month clinic visit for the treatment arm subjects.

Group I: Control Arm- No intervention. Subjects will receive cognitive and lab testing and continue with current management of their cognitive impairment.

Group II: Treatment Arm- In the outpatient setting, one chewable tablet multivitamin (Zn and folic acid containing) plus a titrated dosing of L-histidine powder or capsules starting at 2g consumed before noon escalating every 2 weeks up to 4, 6, then 8 g per day as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* >49 years
* Live at home currently
* Clinical Dementia Score of 3.0 or higher

Exclusion Criteria:

* psychiatric

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating | 12 months
  The median change in the score at 12 months on the Clinical Dementia Rating-Sum of Boxes (CDR-SB; range, 0 to 18, with higher scores indicating greater impairment) between groups looking for regression to higher levels of cognition or conversion to more severe dementia

SECONDARY OUTCOMES:
Histidine blood levels | 3 months
  the comparison in histidine and histamine levels between groups at baseline and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Wells Reynolds, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States